CLINICAL TRIAL: NCT02893891
Title: Metabolic Changes of Fat and Bone Tissue After Radical Bariatric Surgery
Brief Title: Metabolic Changes After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other); Vitkovice Hospital, Ostrava, Czech Republic (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LFOU-SGS-Bariatric Surgery; SGS10/LF/2012 (Other Grant/Funding Number: Medical Faculty, Ostrava University)
Record Dates: First submitted 2016-02-24; First posted 2016-09-09 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-03

CONDITIONS: Grade III Obesity; Type 2 Diabetes Mellitus
Keywords: Obesity; Bariatric medicine; Sleeve gastric resection; Gastric plication; Intragastric ballon; Body composition; Adipokines; Ghrelin; Bone mineral density; Quality of life
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Laparoscopic sleeve gastrectomy (Active Comparator): Patients undergoing bariatric surgery procedure of laparoscopic sleeve gastrectomy.
  Interventions: Procedure: Laparoscopic sleeve gastrectomy
- Laparoscopic gastric plication (Active Comparator): Patients undergoing bariatric surgery procedure of laparoscopic gastric plication.
  Interventions: Procedure: Laparoscopic gastric plication
- Intragastric balloon (Active Comparator): Patients undergoing bariatric surgery procedure with intragastric balloon implantation.
  Interventions: Procedure: Intragastric balloon; Device: Intragastric balloon implantation

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Sleeve gastrectomy involves removing most of the stomach, limiting the amount of food the patient can eat.
  Arms: Laparoscopic sleeve gastrectomy
Procedure: Laparoscopic gastric plication — Laparoscopic gastric plication involves sewing one or more large folds in the stomach. During the laparoscopic gastric plication, the stomach volume is reduced about 70%, which makes the stomach able to hold less and helps the patient eat less.
  Arms: Laparoscopic gastric plication
Procedure: Intragastric balloon — The introduction of the balloon is non-invasive as it is inserted endoscopically (down the oesophagus). The balloon is then filled inside the stomach with a dyed physiological solution, which reduces the volume of the stomach.
  Arms: Intragastric balloon
Device: Intragastric balloon implantation — Intragastric balloons (End-Ball, Medsil) will be implanted in the patients with morbid obesity.
  Arms: Intragastric balloon

SUMMARY:
Literature data clearly demonstrate that treatment of obese patients is very expensive, long and achieve weight loss may not be permanent, and regardless of whether the treatment dominated diet therapy, physical activity, or pharmacotherapy. Experience of the last decade has shown that after surgical interventional treatment of obesity occurs not only long-term (10 years and over) weight loss of 35-40%, but also an important endocrine changes.

In recent years, it was discovered a number of signaling molecules produced by adipose tissue, whose physiological significance beyond the general metabolic aspects organism. The fat is therefore currently understood as an endocrine organ whose hormones modulate the function of many systems, including the skeleton. These hormones include the adipokines that modulate metabolism skeleton as at tissue level (Leptin, Adiponectin) and indirectly - by activation of neurohumoral hypothalamic centers - Leptin.

Studying endocrine interactions between adipose tissue and bone is a highly topical issue. This mutual communication is a homeostatic feedback system in which adipokines and molecules secreted by osteoblasts and osteoclasts are the connecting link active axes fat - bone tissue. However, the mechanisms of this axis remain largely unknown.

DETAILED DESCRIPTION:
Obesity is an important medical problem. The number of obese individuals is increasing continuously in response to various environmental and genetic factors. For some morbidly obese patients, surgery is the only effective type of therapy. Despite bariatric surgery having good outcomes in terms of weight loss, it is associated with some adverse effects: several studies have reported subsequent alterations in bone metabolism. Of the surgical techniques available (laparoscopic gastric banding, Roux-en-Y bypass, biliopancreatic diversion), laparoscopic sleeve gastrectomy (LSG) is currently the technique of choice. Because restrictive procedures such as LSG do not involve bypassing segments of small bowel where micronutrient absorption takes place, fewer metabolic disturbances are expected than with other surgical techniques.

The observed changes in bone metabolism and status in post-bariatric surgery patients potentially involve several mechanisms, including reduced absorption of essential nutrients, diminished calcium absorption leading to secondary hyperparathyroidism, poor vitamin D absorption and restricted energy delivery. In addition, body weight protects against osteoporosis via the bone-strengthening effects of long-term weight bearing. However, long-term decreases in bone mineral density in patients who have undergone successful bariatric surgery are an unexpected, negative effect of this type of therapy.

In the study, parameters of fat and bone tissue and body composition changes are assessed in groups of bariatric patients after LSG, gastric plication and intragastric balloon treatment. Other anticipated benefits of the study treatment include improving the quality of life of. lt will also lead to the introduction of new processes, materials and methods. lt is also possible to expect shortening of the hospital stay, decrease in postoperative morbidity, and the possibility to perform the procedure on an outpatient basis.

The study has been designed as a prospective study, which is in conformity with the principles and guidelines of the Helsinki Declaration, good clinical practice and has been approved by the Ethical Committee of the Faculty of Medicine, University of Ostrava.

The patients enrolled in the study are followed for the period of twelve months. Timetable of the study procedures and controls:

Preoperative examination:

* Demographic data on age, sex, weight, height, smoking
* Assessment of body composition and sampling of blood
* Questionnaires for quality of Life Examination 3 months postoperatively
* Assessment of body composition and sampling of blood
* Questionnaires for quality of Life Examination 6 months after surgery
* Assessment of body composition and sampling of blood
* Questionnaires for quality of Life Examination 12 months after surgery
* Assessment of body composition and sampling of blood
* Questionnaires for quality of Life

Statistical data processing for statistical evaluation descriptive statistics are used (arithmetical average, standard deflection, frequency tables), X2 test, Fisher's exact test, analysis of variance (ANOVA), calculating of the OR (odds ratio) with 95 % confidence intervals, and logistic regression. Statistical tests are evaluated at the significance level of 5%. Statistical analysis is performed in the "Stata 10" programme. Program EpiData is used for data collection.

ELIGIBILITY:
Inclusion Criteria:

* History of conservative obesity treatments selected according to criteria IFSO (BMI greater than 40 or greater than 35 with comorbidities)

Exclusion Criteria:

* Thyroid disease
* Diseases of the digestive system associated with disorders of intestinal absorption
* History of corticosteroid therapy in the past 12 months

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in serum levels of adipose tissue hormones | 18 months
  To analyze the dynamics of changes in serum levels of adipose tissue hormones (Leptin, Adiponectin) in adults after bariatric treatment of malignant obesity (BMI> 35). Points of measurements: before the planned intervention and then in intervals of 3, 6, 12, and 18 months after procedure.
Changes in serum levels of lipids | 18 months
  To analyze the dynamics of changes in serum levels of lipids in adults after bariatric treatment of malignant obesity (BMI> 35). In the study, serum concentrations of the following lipids will be measured: tricylglycerols, total cholesterol, high-density lipoprotein, low-density lipoprotein cholesterol, Apo D and Apo E. The measurements will be performed before the planned intervention and then in intervals at 3, 6, 12, and 18 months after the procedure. The results will be presented in respective units (mmol/L, mg/dL, etc.).
Changes in serum levels of osteomarkers | 18 months
  To analyze the dynamics of changes in serum levels of usual panel of osteomarkers in adults after bariatric treatment of malignant obesity (BMI> 35). The following serum levels markers of bone resorption and formation will be assessed: CTx, P1NP, ALP, RANKL, FGF 23, Osteocalcin, Osteopontin and vitamin D2 and D3. The measurements will be performed before the planned intervention and then in intervals at 3, 6, 12, and 18 months after the procedure. The results will be presented in respective units (mmol/L, mg/dL, etc.).
IWQOL Questionnaire evaluation | 18 months
  Evaluation of effects of different types of bariatric interventions on quality of life will be performed by using the IWQOL questionnaire. Improvement from baseline quality of life as measured by standardized IWQOL patient questionnaire (http://www.qualityoflifeconsulting.com/iwqol-lite.html) intended to measure the patient health status.
SF-36 Questionnaire evaluation | 18 months
  Evaluation of effects of different types of bariatric interventions on quality of life will be performed using the SF-36 questionnaire. Improvement from baseline quality of life as measured by standardized SF-36 patient questionnaire intended to measure the patient health status.

SECONDARY OUTCOMES:
Long-term weight reduction assessment in kgs | 18 months
  Evaluation of the success of treatment in terms of long-term weight reduction (difference in body weight in kilograms at the beginning vs. the end of the observation period of 18 months), expressed as TBL (total body weight loss), EWL (excess weight loss), and EBL (excess BMI loss).
Effectiveness evaluation | 18 months
  Evaluation of the effectiveness of the specified bariatric procedures, including new intragastric balloons. The following parameters will be assessed at 3, 6, and 12 months: 1) Per cent total body weight loss and excess weight loss at 12 months, 2) Changes in fasting glycaemia, insulin and hemoglobin A1C at 12 months; 3) Reduction in diabetes medication requirements (for diabetic cohort) at 12 months, and 4) Occurrence rate of serious adverse events judged to be probably or definitely related to the study device.

CONTACTS AND LOCATIONS:
Overall Officials: Marek Bužga, MSc., Ph.D., Principal Investigator — Faculty of Medicine, Ostrava University, Ostrava
Locations (2):
- Czechia (2):
  - Vítkovice Hospital Ostrava, Ostrava, Moravian-Silesian Region
  - University Hospital Ostrava, Ostrava, Moravian-Silesian Region

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Background] Suter M, Calmes JM, Paroz A, Giusti V. A 10-year experience with laparoscopic gastric banding for morbid obesity: high long-term complication and failure rates. Obes Surg. 2006 Jul;16(7):829-35. doi: 10.1381/096089206777822359. PMID 16839478
- [Background] Bose M, Olivan B, Teixeira J, Pi-Sunyer FX, Laferrere B. Do Incretins play a role in the remission of type 2 diabetes after gastric bypass surgery: What are the evidence? Obes Surg. 2009 Feb;19(2):217-229. doi: 10.1007/s11695-008-9696-3. Epub 2008 Sep 27. PMID 18820978
- [Background] Buchwald H, Oien DM. Metabolic/bariatric surgery Worldwide 2008. Obes Surg. 2009 Dec;19(12):1605-11. doi: 10.1007/s11695-009-0014-5. PMID 19885707
- [Background] Koerner A, Kratzsch J, Kiess W. Adipocytokines: leptin--the classical, resistin--the controversical, adiponectin--the promising, and more to come. Best Pract Res Clin Endocrinol Metab. 2005 Dec;19(4):525-46. doi: 10.1016/j.beem.2005.07.008. PMID 16311215
- [Background] Magni P, Dozio E, Galliera E, Ruscica M, Corsi MM. Molecular aspects of adipokine-bone interactions. Curr Mol Med. 2010 Aug;10(6):522-32. doi: 10.2174/1566524011009060522. PMID 20642443
- [Background] Pobeha P, Ukropec J, Skyba P, Ukropcova B, Joppa P, Kurdiova T, Javorsky M, Klimes I, Tkac I, Gasperikova D, Tkacova R. Relationship between osteoporosis and adipose tissue leptin and osteoprotegerin in patients with chronic obstructive pulmonary disease. Bone. 2011 May 1;48(5):1008-14. doi: 10.1016/j.bone.2011.02.017. Epub 2011 Mar 1. PMID 21376149
- [Background] Boyce BF, Xing L. Functions of RANKL/RANK/OPG in bone modeling and remodeling. Arch Biochem Biophys. 2008 May 15;473(2):139-46. doi: 10.1016/j.abb.2008.03.018. Epub 2008 Mar 25. PMID 18395508
- [Background] Makovey J, Naganathan V, Seibel M, Sambrook P. Gender differences in plasma ghrelin and its relations to body composition and bone - an opposite-sex twin study. Clin Endocrinol (Oxf). 2007 Apr;66(4):530-7. doi: 10.1111/j.1365-2265.2007.02768.x. PMID 17371471
- [Background] Hamrick MW, Ferrari SL. Leptin and the sympathetic connection of fat to bone. Osteoporos Int. 2008 Jul;19(7):905-12. doi: 10.1007/s00198-007-0487-9. Epub 2007 Oct 9. PMID 17924050
- [Background] Gomez-Ambrosi J, Rodriguez A, Catalan V, Fruhbeck G. The bone-adipose axis in obesity and weight loss. Obes Surg. 2008 Sep;18(9):1134-43. doi: 10.1007/s11695-008-9548-1. Epub 2008 Jun 19. PMID 18563500
- [Background] Greco EA, Fornari R, Rossi F, Santiemma V, Prossomariti G, Annoscia C, Aversa A, Brama M, Marini M, Donini LM, Spera G, Lenzi A, Lubrano C, Migliaccio S. Is obesity protective for osteoporosis? Evaluation of bone mineral density in individuals with high body mass index. Int J Clin Pract. 2010 May;64(6):817-20. doi: 10.1111/j.1742-1241.2009.02301.x. PMID 20518955
- [Background] Wucher H, Ciangura C, Poitou C, Czernichow S. Effects of weight loss on bone status after bariatric surgery: association between adipokines and bone markers. Obes Surg. 2008 Jan;18(1):58-65. doi: 10.1007/s11695-007-9258-0. Epub 2007 Dec 11. PMID 18074189
- [Derived] Buzga M, Svagera Z, Tomaskova H, Hauptman K, Holeczy P. Metabolic Effects of Sleeve Gastrectomy and Laparoscopic Greater Curvature Plication: an 18-Month Prospective, Observational, Open-Label Study. Obes Surg. 2017 Dec;27(12):3258-3266. doi: 10.1007/s11695-017-2779-2. PMID 28674838